CLINICAL TRIAL: NCT06755697
Title: Comparative Efficacy of Intra-articular vs. MRI-guided Extra-articular Dextrose Injections in Knee Osteoarthritis Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin-Fen Hsieh, Study Principal Investigator, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20240717R
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis; Glucose; Prolotherapy; MRI; Physical Therapy; Rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-articular US-guided hypertonic dextrose injection, IA group (Active Comparator): IA injection: 5 ml of 20% dextrose (2ml vitagen in 2ml normal saline and 1ml 1% xylocain) will be injected. The ultrasound transducer (L18-4, Philips EPI Q5) is placed transversely over the patient's suprapatellar pouch while the patient lies supine with the knee actively extended and ankle dorsiflexed. The injectate will be injected into the suprapatellar pouch via transverse view, in-plane, lateral-to-medial approach with a 3.8 cm 22-gauge needle under US guidance.
  Physical therapy: The physical therapy program includes physical modalities (heat therapy and electric therapy) and therapeutic exercise (stretching, ROM exercise, and strengthening), three times a week, and will be continued for 4 weeks.
  Interventions: Other: Intra-articular US-guided hypertonic dextrose injection, IA group
- Extra-articular US-guided injection targeting MRI-positive lesion sites, EA group. (Active Comparator): Patients in the EA group will receive MRI examination of the knee without contrast.
  Detailed physical examinations (PE) will also be done for each subject. The PEs include inspection, palpation for local tenderness and crepitus, signs of effusion, assessment of range of motion, provocative meniscal testing, and ligamentous tests for laxity. (16) A total of 5 ml of 20% dextrose (2ml vitagen in 2ml normal saline and 1ml 1% xylocain) will be injected to the target areas which has been shown abnormal on MRI images with a 3.8 cm 22-gauge needle under US guidance. For lesions of the deep structures or bone marrow lesion, a 7-cm 23 or 21 gauge needles may be used. Same as the IA group, EA hypertonic dextrose injection will be done at the 0, 2nd, and 4th weeks, as well as physical therapy during the first 4 weeks.
  Interventions: Other: Extra-articular US-guided injection targeting MRI-positive lesion sites, EA group.

INTERVENTIONS:
Other: Intra-articular US-guided hypertonic dextrose injection, IA group — IA injection: 5 ml of 20% dextrose (2ml vitagen in 2ml normal saline and 1ml 1% xylocain) will be injected. The ultrasound transducer (L18-4, Philips EPI Q5) is placed transversely over the patient's suprapatellar pouch while the patient lies supine with the knee actively extended and ankle dorsiflexed. The injectate will be injected into the suprapatellar pouch via transverse view, in-plane, lateral-to-medial approach with a 3.8 cm 22-gauge needle under US guidance.
  Physical therapy: The physical therapy program includes physical modalities (heat therapy and electric therapy) and therapeutic exercise (stretching, ROM exercise, and strengthening), three times a week, and will be continued for 4 weeks.
  Arms: Intra-articular US-guided hypertonic dextrose injection, IA group
Other: Extra-articular US-guided injection targeting MRI-positive lesion sites, EA group. — Patients in the EA group will receive MRI examination of the knee without contrast. Detailed physical examinations (PE) will also be done for each subject. The PEs include inspection, palpation for local tenderness and crepitus, signs of effusion, assessment of range of motion, provocative meniscal testing, and ligamentous tests for laxity. A total of 5 ml of 20% dextrose (2ml vitagen in 2ml normal saline and 1ml 1% xylocain) will be injected to the target areas which has been shown abnormal on MRI images with a 3.8 cm 22-gauge needle under US guidance. For lesions of the deep structures or bone marrow lesion, a 7-cm 23 or 21 gauge needles may be used. Same as the IA group, EA hypertonic dextrose injection will be done at the 0, 2nd, and 4th weeks, as well as physical therapy during the first 4 weeks.
  Arms: Extra-articular US-guided injection targeting MRI-positive lesion sites, EA group.

SUMMARY:
Osteoarthritis (OA) is a serious worldwide public health concern, causing increased disability-adjusted life years (DALY), the reasons of which include rising prevalence of obesity and increasing older populations. The knee is one of the most easily injured joint in the body, and knee OA can become a chronic and disabling condition that pose a threat to not only the patient but also his or her caretakers and healthcare resources. The prevalence of knee OA is 5% - 15% in men over 60 years, and 10% - 25% in women aged more than 60.

Knee OA can result from injuries, diseases, or wear and tear from overuse. It refers to structural changes that affect subchondral bone, articular cartilage, menisci, ligaments, synovium, and other joint structures. Currently, there are several conservative management of knee OA, including physiotherapy (therapeutic exercise, diathermy, electrotherapy), oral or topical medications, intra-articular and extra-articular injections, and radiofrequency.

There are various substances used in injections for knee OA, among which are corticosteroid, platelet-rich plasma (PRP), AmnioFix, exosome, dextrose, and hyaluronic acid (HA). Compared with PRP, AmnioFix, exosome, and HA, which are not covered by the health insurance system, dextrose is a readily available and cost-effective substance. The principle of hypertonic dextrose injection, "prolotherapy", is injection of small volumes of the irritant solution at or around the lesion in order to stimulate fibroblast and vascular proliferation, local tissue healing, reduction of joint instability, thus resulting in pain relief. Previous studies have demonstrated that prolotherapy resulted in clinically meaningful sustained improvement of function and pain in knee OA, and there were no severe adverse events related to hypertonic dextrose injection. A study in 2023 showed that among various dextrose concentrations, higher concentrations demonstrated greater improvement of knee OA, thus 20% dextrose is recommended.

Regarding the site of dextrose injection in knee OA, previous studies demonstrated comparable effects of intra-articular and extra-articular injections. The periarticular injections include points around the knee where periarticular nerves exit the joint capsule, and acupuncture points at upper medial and lateral parts of knee joint. A study in 2024 revealed that prolotherapy combining intra-articular with peri-articular perineural injection resulted in better pain alleviation and improvement in knee joint function in knee OA. There are several choices of imaging modality for recognizing the sites of lesion in knee OA, such as X-ray, ultrasound (US), and magnetic resonance imaging (MRI). Radiography is used to assess osteophytes, joint space narrowing, and subchondral sclerosis, but it has limited ability to detect synovial inflammation, joint effusion, soft tissue abnormalities, and early cartilage damage. US can be used to evaluate synovial fluid and cartilage thickness, but not deep structures (e.g. subchondral bone change, meniscus tear, and ACL tear, etc.). On the other hand, MRI is an optimal and accurate imaging choice for visualizing soft tissue as well as deep structures (e.g. ACL, meniscus, etc) in knee OA. The MRI findings of knee OA includes cartilage damage, meniscus tear, bone marrow lesions, synovitis, ligamentous laxity, and osteophytes. The detection of bony lesions can aid intraosseous Infiltrations, and signs of ligamentous laxity also provides target for ligaments injection. However, there is no current evidence on the effectiveness of prolotherapy targeting knee OA lesion sites according to MRI findings.

Because the effectiveness of prolotherapy targeting lesion sites according to MRI findings has not been well established, the investigators aim to investigate whether injecting dextrose into MRI-positive lesion sites is more beneficial for knee OA comparing to intra-articular injections. The investigators hypothesize that MRI could be a good choice for the guidance of prolotherapy targets.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a serious worldwide public health concern, and there are several conservative management of knee OA. Evidence showed that intra-articular and extra-articular injections are beneficial for knee OA. Compared with PRP, AmnioFix, exosome, and HA, which are not covered by the health insurance system, dextrose is a readily available and cost-effective substance. There are several choices of imaging modality for recognizing the sites of lesion in knee OA, such as X-ray, ultrasound (US), and magnetic resonance imaging (MRI). MRI is an optimal and accurate imaging choice for visualizing soft tissue as well as deep structures. The MRI findings of knee OA includes cartilage damage, meniscus tear, bone marrow lesions, synovitis, ligamentous lesions, and osteophytes. The detection of bony lesions can aid intraosseous Infiltrations. However, there is no current evidence on the effectiveness of prolotherapy targeting knee OA lesion sites according to MRI findings. Thus, the investigators aim to investigate whether injecting dextrose into MRI-positive lesion sites is more beneficial for knee OA comparing to intra-articular injections.

ELIGIBILITY:
Inclusion Criteria:

1. . age between 45 to 80 years old;
2. . meet at least three of the six American College of Rheumatology (ACR) criteria, including age over 50 years, morning stiffness less than 30 minutes, crepitus in passive knee movements, bony tenderness, bony enlargement, and no palpable warmth;
3. . radiologic grading of 2 or 3 according to Kellgren-Lawrence criteria;
4. showing willingness to receive prolotherapy.

Exclusion Criteria:

1. . severe systemic disorders including cancer, uncontrolled diabetes mellitus, sepsis, or cardiopulmonary diseases;
2. . history of anticoagulation therapy, knee injection over the past three months;
3. . history of knee surgery or candidates for knee arthroplasty;
4. . history of drug abuse;
5. . a history of intolerance to prolotherapy;
6. . pregnancy;
7. . infectious arthritis, inflammatory joint diseases, joint dysplasia;
8. Body Mass Index (BMI) greater than 35 kg/m2;
9. . not suitable or no willing to received MRI examination of the knee.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The Western Ontario McMaster University Osteoarthritis Index（WOMAC） | Change between baseline and at 1.5 months, 3 months, 6 months after the beginning of the treatment.
  The WOMAC is a questionnaire evaluating the severity of osteoarthritis using pain, stiffness, and function subscales. The WOMAC composite score is constructed as the weighted average of the 3 subscale scores, and it ranges from 0 (worst) to 100 (best) for depicting knee-related quality-of-life. For WOMAC, the minimal clinical important difference (MCID) for knee OA has been reported as a change of 12 points on a 0- to 100-mm visual analog scale. According to previous studies, WOMAC is responsive to clinical changes.

SECONDARY OUTCOMES:
The pain visual analog scale (VAS) | Change between baseline and at 1.5 months, 3 months, 6 months after the beginning of the treatment.
  The pain VAS is obtained using a 100-mm-long horizontal line, with 0 mm on the left, indicating no pain, and 100 mm on the right, indicating very severe pain. The MCID of pain VAS for knee OA ranged from 10 to 19.9 points, according to previous studies.
The 36-item Short Form Health Survey (SF-36) | Change between baseline and at 1.5 months, 3 months, 6 months after the beginning of the treatment.
  The general health status and quality of life will be measured with the SF-36. The SF-36 is composed of 8 subscales including the following components: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each subscale generates a score ranging from 0 to 100, and higher scores indicate better quality of life. A Chinese-language version will be used for which the psychometric properties have been established.
Timed Up and Go (TUG) test | Change between baseline and at 1.5 months, 3 months, 6 months after the beginning of the treatment.
  TUG test is a measure of dynamic balance which has good inter-rater and test-retest reliability. During a TUG test, it is timed when a patient rises from a chair, walks 3 meters, turns and walks back, and then sits down again. The MCID of TUG test has been reported as 3.4 seconds in patients with lumbar stenosis.
Self-assessment of the treatment effect | Change between baseline and at 1.5 months, 3 months, 6 months after the beginning of the treatment.
  Self-assessment of the treatment effect: Patient's evaluation of the treatment effect consists of the answer to one question: "Is the treatment effective?" scored on a Likert scale (very effective=5, effective=4, same=3, worse=2, much worse=1). (This item is not evaluated at baseline.)

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan